CLINICAL TRIAL: NCT04093115
Title: A Clinical Trial to Evaluate the Efficacy and Safety of CX1106 in Patients With Metastatic/Recurrent Head and Neck Squamous Cell Carcinoma After Failure of or Unfit for Platinum-containing Therapy
Brief Title: Study of CX1106 in Patients With Advanced Head and Neck Squamous Cell Carcinoma
Acronym: HNSCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated voluntarily by the sponsor due to changes in clinical development strategy.
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC-DIAO-004
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CX1106 (Experimental): CX1106 740 mg/m2 as a 24-hour continuous infusion for 5 days every 3 weeks (3 weeks/cycle, 4-6 cycles)
  Interventions: Drug: CX1106

INTERVENTIONS:
Drug: CX1106 — administration of CX1106 at 740 mg/m2 as a 24-hour continuous infusion for 5 days (120 h, d1-5), 21 days per cycle, no more than 6 cycles

SUMMARY:
CX1106 is a novel inhibitor of thymidylate synthase (TS) developed as a potential antitumor agent by virtue of the rate limiting role of TS in the biosynthesis of thymidine. CX1106 differs from other TS inhibitors such as pemetrexed, raltitrexed, CB3717, and fluorouracil in that it does not require active transport for uptake into cells. CX1106 also lacks a glutamate moiety and thus does not require polyglutamation for antitumor activity. More than 1000 patients with various malignancies have been treated with CX1106 to date in previous various clinical trials.

The investigators suggest a study of CX1106 in patients with recurrent or metastatic HNSCC who are resistant or ineligible/intolerant to platinum-based chemotherapy. The aim of current trial is to evaluate the antitumor efficacy and safety profile of CX1106.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HNSCC (excluding nasopharyngeal carcinoma);
* At least one measurable lesion (spiral CT scan long diameter ≥ 10 mm or enlarged lymph node short diameter ≥ 15 mm by RECIST 1.1);
* Documented disease progression after prior platinum-based systematic therapy; or prior platinum-based adjuvant/neoadjuvant therapy with documented disease progression within 24 weeks after treatment completion;
* Expected overall survival≥ 3 months;
* ECOG PS≤1;

Exclusion Criteria:

•Hematologic, renal, and hepatic function as defined below:

Absolute neutrophil count (ANC) <1.5×109 /L or platelet <100×109 /L or hemoglobin <9 g/dL; Total bilirubin >1.5×the upper limit of normal range(ULN); Aspartate aminotransferase (AST) and/or Alanine transaminase (ALT) and/or Alkaline phosphatase (ALP) >1.5×ULN without liver metastases ; AST and/or ALT and/or ALP levels >5×ULN with liver metastases. Primary hepatocellular carcinoma: Child-Pugh liver is grade C; Serum creatinine>1.5 ×ULN or creatinine clearance (CL) < 60 mL/min; International normalized ratio (INR) or activated partial thromboplastin time (aPPT) >1.5×ULN;

* Patients who has accepted systemic anti-tumor therapy, including chemotherapy, radiotherapy, hormonal therapy , biologics therapy or immunotherapy within 4 weeks;
* Any unresolved Grade ≥2 toxicity by NCI CTCAE 5.0 from previous anticancer therapy excluding skin pigmentation and alopecia;
* Untreated brain metastases or symptoms of brain metastases cannot be controlled more than 4 weeks;
* Other kinds of malignancies [excluding stage IB or lower grade cervical cancer，noninvasive basal cell or squamous cell cancer, breast cancer with complete remission (CR) > 10 years ,melanoma with CR >10 years or other malignant tumors with CR > 5 years];
* Any of the following gastrointestinal disease:

Need intravenous nutrition; Received treatment for active peptic ulcer disease in the past 6 months; Active gastrointestinal bleeding unrelated to cancer in the past 3 months; Persistent 3 or 4 grade chronic diarrhea although with treatment;

* Presence of hemorrhage (hemoptysis) , thrombosis，or currently receiving treatment with warfarin, aspirin, low molecular weight heparin (LMWH), or any other anti-platelet drugs(low dose of abovementioned drugs for prophylaxis are allowed);
* Active infections, mental and neurological diseases;
* Prior to enrollment within 12 months , patients who had cardiovascular and cerebrovascular disease, deep vein thrombosis or pulmonary embolism within 6 months; or uncontrolled hypertension,systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg;
* Prior to enrollment within 30 days , patients who had Major surgical procedure, open biopsy, or significant traumatic injury;
* Hepatitis B surface antigen (HBsAg) positive and HBV-DNA≥ 2000 IU / mL;hepatitis C virus (HCV) antibody positive; and cirrhosis;
* Known history of human immunodeficiency virus (HIV) infection;
* Pregnant or lactating women or those who do not take contraceptives, including men;
* Prior to enrollment within 30 days , patients who have participated in other clinical trials of anti-tumor medicine;
* Diseases which would severely endanger the security of patients or influence the completion of this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  Defined as the percentage of subjects with confirmed complete response (CR) or partial response (PR) according to the Response Evaluation in Solid Tumor Criteria 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 24 months
  Defined as the proportion of patients with confirmed complete response, partial response, and stable disease (CR + PR + SD) according to the Response Evaluation in Solid Tumor Criteria 1.1 (RECIST 1.1)
Progression-free survival (PFS) | up to 24 months
  Defined as the duration time from the first CX1106 administration to confirmed disease progression (PD) or death of any reason, whichever occurred first
Safety profile as assessed by the incidence, duration, and severity of adverse events | up to 24 months
  Incidence, duration, and severity of AEs measured by laboratory assessments and physical findings according to NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: YuanKai Shi, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science

IPD SHARING:
Plan to Share IPD: No